CLINICAL TRIAL: NCT06702566
Title: The Significance of Serum Ferritin in the Diagnosis, Differential Diagnosis, and Prognosis of Immune-related Adverse Event (irAE)
Brief Title: The Effect of Serum Ferritin in irAE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: E20240619
Record Dates: First submitted 2024-07-16; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-07

CONDITIONS: Immune-related Adverse Event; Malignant Solid Tumors; Acute Leukemia; Serum Ferritin
MeSH Terms: interventions — Immune Checkpoint Inhibitors; Antineoplastic Agents

STUDY DESIGN:
Intervention Model Description: This is a prospective clinical study to clarify serum ferritin as a biomarker for the diagnosis, differential diagnosis and prognosis of immune-related adverse event(irAE). A total of 1500 patients with definitive diagnosis of malignant solid tumor or acute leukemia will be enrolled in this study. Patients are divided into 3 groups according to the anti-tumor therapy they are to receive. Three groups will be set up, namely group A: immunotherapy group (patients will be treated with immunotherapy, or immuno- plus targeted therapy, or immuno- plus chemotherapy); group B: targeted therapy group (patients will be treated with targeted monotherapy, targeted plus chemotherapy); group C: chemotherapy group (patients will be treated with chemotherapy).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A: Serum ferritin in patients receiving immunotherapy (Experimental): Patients will receive standardized anti-tumor therapy including immunotherapy according to clinical guidelines. Patients who treated with immuno-monotherapy, or immuno- plus targeted therapy, or immuno- plus chemotherapy will be recruit in to test the serum ferritin level
  Interventions: Drug: PD-1 and PD-L1 inhibitor; Drug: Targeted drugs; Drug: chemotherapy drugs
- B: Serum ferritin in patients receiving targeted therapy (Active Comparator): Patients will receive standardized anti-tumor therapy including targeted therapy according to clinical guidelines. Patients who treated with targeted monotherapy, or targeted plus chemotherapy will be recruit in to test the serum ferritin level
  Interventions: Drug: Targeted drugs; Drug: chemotherapy drugs
- C: Serum ferritin in patients receiving chemotherapy (Active Comparator): Patients will receive standardized anti-tumor therapy including chemotherapy according to clinical guidelines. Patients who treated with chemotherapy will be recruit in to test the serum ferritin level
  Interventions: Drug: chemotherapy drugs

INTERVENTIONS:
Drug: PD-1 and PD-L1 inhibitor — PD-1 inhibitor includes pembrolizumab，Nivolumab，Sintilimab，tislelizumab，Triplimab，Camrelizumab, Serplulimab.
  PD-L1 inhibitor includes durvalumab,Atezolizumab,Adebrelimab,Envafolimab.
  Arms: A: Serum ferritin in patients receiving immunotherapy
Drug: Targeted drugs — Targeted drugs includes EGFR-TKIs,ALK-TKIs,Multitargeted Tyrosine Kinase Inhibitors, VEGF antibody, EGFR antibody, antibody-drug conjugates drugs
  Arms: A: Serum ferritin in patients receiving immunotherapy; B: Serum ferritin in patients receiving targeted therapy
Drug: chemotherapy drugs — Chemotherapy drugs are determined based on the investigator's decision.

SUMMARY:
This is a prospective clinical study to clarify serum ferritin as a biomarker for the diagnosis, differential diagnosis and prognosis of immune-related adverse event(irAE).

DETAILED DESCRIPTION:
A total of 1500 patients with definitive diagnosis of malignant solid tumor or acute leukemia will be enrolled in this study. Patients are divided into 3 groups according to the anti-tumor therapy they are to receive. Three groups will be set up, namely group A: immunotherapy group (patients will be treated with immunotherapy, or immuno- plus targeted therapy, or immuno- plus chemotherapy); group B: targeted therapy group (patients will be treated with targeted monotherapy, targeted plus chemotherapy); group C: chemotherapy group (patients will be treated with chemotherapy). All patients received blood biochemistry and imaging at baseline, and adverse events were monitored. If a patient in the immunotherapy group presents with an AE, the AE is diagnosed by a multi-disciplinary MDT team including oncologists, rheumatologists, immunologists, respiratory pathologists, radiologists, and pathologists, and further diagnosed as irAE or non-irAE. All patients underwent hematologic testing every 3 days (at least 3 times) after the onset of AE including: blood routine examination, ferritin, CRP, D-dimer, and cytokines (IL-1β, IL-6, and TNF-α)until recovery from AE. Patients without AE will re-testing of baseline blood biochemistry every 4 treatment cycles.

ELIGIBILITY:
Inclusion Criteria:

Only patient who meet all the following conditions can be selected for this trial:

1. Patients voluntarily sign informed consent;
2. The age was 18-75 years old, and the gender was not limited;
3. Patients with definitive diagnosis of malignant solid tumor or acute leukemia;
4. Patients enrolled in will be treated with immunotherapy (including immuno- monotherapy，or immuno- plus targeted therapy, or immuno- plus chemotherapy), or targeted therapy (including targeted monotherapy, or targeted plus chemotherapy), or chemotherapy.
5. The Eastern Cooperative Oncology Group (ECOG) scored 0 or 1 or 2 for physical fitness;
6. Sufficient bone marrow reserve at screening, defined as:

   * Neutrophil absolute value (ANC) > 1.5 × 10^9/L；
   * Lymphocyte absolute value (ALC) ≥ 0.3 × 10^9/L；
   * Platelet (PLT) ≥ 100 × 10^9/L；
   * Hemoglobin (HGB) ≥ 100g / L;
7. The screening has appropriate organ function and meets the following criteria:

   * Aspartate aminotransferase (AST) ≤ 2.5 times ULN (due to tumor infiltration ≤ 5 times ULN);
   * Alanine aminotransferase (ALT) ≤ 2.5 times ULN (due to tumor infiltration ≤ 5 times ULN);
   * Total serum bilirubin ≤ 1.5 times ULN (due to tumor infiltration ≤ 3 times ULN);
   * Serum creatinine (SCR) ≤ 1.5 times ULN, or creatinine clearance rate ≥ 60ml / min;
   * Have the lowest level of lung reserve, defined as ≤ grade 1 dyspnea and oxygen saturation > 91% in non oxygen breathing state;
   * International normalized ratio (INR) ≤ 1.5 times ULN, and activated partial prothrombin time (APTT) ≤ 1.5 times ULN;
8. The urine pregnancy test of women of childbearing age is negative. Any male and female patient with fertility must agree to use effective contraceptive methods during the whole study and at least 1 year after the study treatment.

Exclusion Criteria:

Patient who meet any of the following conditions well excluded in this trial:

1. Active systemic autoimmune disease is known before screening and is under treatment;
2. Those who stopped systemic hormone therapy for less than 2 weeks before enrollment；
3. Those who have received organ / tissue transplantation before screening;
4. Those who meet any of the following conditions during screening:

   * positive for hepatitis B surface antigen (HBsAg) and / or hepatitis B e antigen (HBeAg);
   * hepatitis B e antibody (HBE AB) and / or hepatitis B core antibody (HBC AB) are positive, and the copy number of HBV-DNA is greater than the lower measurable limit;
   * positive for hepatitis C antibody (HCV AB);
   * positive anti Treponema pallidum antibody (TP AB);
   * HIV antibody test positive;
   * the copy number of EBV-DNA and cmv-dna is greater than the lower measurable limit;
5. The heart meets any of the following conditions during screening:

   * left ventricular ejection fraction (LVEF) ≤ 50% (echo);
   * New York Heart Association (NYHA) class III or IV congestive heart failure;
   * hypertension (systolic blood pressure ≥ 140mmHg and / or diastolic blood pressure ≥ 90mmHg) or pulmonary hypertension that has not been controlled by standard treatment;
   * have had myocardial infarction or cardiac surgery within 12 months before cell transfusion;
   * clinically significant valvular disease.
6. There are clinical emergencies (such as intestinal obstruction or vascular compression) requiring urgent treatment due to tumor body obstruction or compression during screening;
7. Patients with active bleeding during screening;
8. Patients with deep venous thrombosis or pulmonary embolism within 6 months before screening;
9. Those who received live vaccine within 6 weeks before screening;
10. Patients with active infection and need treatment during screening;
11. Poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2024-07-04 (Actual); Primary Completion 2026-07-16 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
calculated cut-off value for serum ferritin in the diagnosis of irAE | 1 year
Determining the sensitivity and specificity of serum ferritin in the diagnosis of irAE | 1 year
Determining baseline level of serum ferritin predicts irAE occurrence | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Xiubao Ren, M.D, Ph.D, Principal Investigator — ianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China